CLINICAL TRIAL: NCT00272792
Title: A Phase 3, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of Phenoptin to Increase Phenylalanine Tolerance in Phenylketonuric Children on a Phenylalanine-restricted Diet
Brief Title: Study of Phenoptin to Increase Phenylalanine Tolerance in Phenylketonuric Children on a Phenylalanine-restricted Diet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKU-006
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Results first posted 2009-07-09 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-07

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

ARMS (2):
- Sapropterin Dihydrochloride (Experimental): Phenoptin, provided in tablets containing 100 mg of sapropterin dihydrochloride each, was administered orally once daily in the morning as the number of tablets equivalent to a 20mg/kg/day dose dissolved in 4-8 oz (120-240 mL) of water or apple juice for 6 weeks. A follow-up call or visit was made 4 weeks later during this double-blind, placebo-controlled study.
  Interventions: Drug: Sapropterin Dihydrochloride
- Placebo (Placebo Comparator): Placebo, provided as tablets similar to Phenoptin tablets, was administered orally once daily in the morning as the number of tablets equivalent to a 20mg/kg/day dose dissolved in 4 8 oz (120-240 mL) of water or apple juice. for 6 weeks. A follow-up call or visit was made 4 weeks later during this double-blind, placebo-controlled study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sapropterin Dihydrochloride — Phenoptin, provided in tablets containing 100 mg of sapropterin dihydrochloride each, was administered orally once daily in the morning as the number of tablets equivalent to a 20mg/kg/day dose dissolved in 4-8 oz (120-240 mL) of water or apple juice for 6 weeks. A follow-up call or visit was made 4 weeks later during this double-blind, placebo-controlled study.
  Arms: Sapropterin Dihydrochloride
Drug: Placebo — Placebo, provided as tablets similar to Phenoptin tablets, was administered orally once daily in the morning as the number of tablets equivalent to a 20mg/kg/day dose dissolved in 4 8 oz (120-240 mL) of water or apple juice. for 6 weeks. A follow-up call or visit was made 4 weeks later during this double-blind, placebo-controlled study.
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to evaluate the ability of Phenoptin to increase phenylalanine (phe) tolerance in children with phenylketonuria who are following a phe-restricted diet.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PKU with hyperphenylalaninemia (HPA) documented by at least one blood Phe measurement >/=360 umol/L (6 mg/dL)
* Under dietary control with a Phe-restricted diet as evidenced by:· Estimated daily Phe tolerance </=1000 mg/day
* At least 6 months of blood Phe control (mean level of </=480 μmol/L) prior to enrolling in the study
* Aged 4 to 12 years inclusive at screening
* A blood Phe level </=480 μmol/L at screening
* Female subjects of childbearing potential (as determined by the principal investigator) must have a negative blood or urine pregnancy test at entry (prior to the first dose). Note: All female subjects of childbearing potential and sexually mature male subjects must be advised to use a medically accepted method of contraception throughout the study. Female subjects of childbearing potential must be willing to undergo periodic pregnancy tests during the course of the study
* Willing and able to comply with all study procedures
* Willing to provide written assent (if applicable) and written informed consent by a parent or legal guardian after the nature of the study has been explained and prior to any research-related procedures

Exclusion Criteria:

* Any condition that, in the view of the PI, renders the subject at high risk from treatment compliance and/or completing the study
* Prior history of organ transplantation
* Perceived to be unreliable or unavailable for study participation or have parents or legal guardians who are perceived to be unreliable or unavailable
* Use of any investigational agent within 30 days prior to screening, or requirement for any investigational agent or vaccine prior to completion of all scheduled study assessments
* ALT > 2 times the upper limit of normal (i.e., Grade 1 or higher based on World Health Organization Toxicity Criteria) at screening
* Concurrent disease or condition that would interfere with study participation or safety (e.g., seizure disorder, oral steroid-dependent asthma or other condition requiring oral or parenteral corticosteroid administration, or insulin-dependent diabetes)

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2006-02; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Los Angeles, California
  - Oakland, California
  - Sacramento, California
  - San Jose, California
  - Chicago, Illinois
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Trefz FK, Burton BK, Longo N, Casanova MM, Gruskin DJ, Dorenbaum A, Kakkis ED, Crombez EA, Grange DK, Harmatz P, Lipson MH, Milanowski A, Randolph LM, Vockley J, Whitley CB, Wolff JA, Bebchuk J, Christ-Schmidt H, Hennermann JB; Sapropterin Study Group. Efficacy of sapropterin dihydrochloride in increasing phenylalanine tolerance in children with phenylketonuria: a phase III, randomized, double-blind, placebo-controlled study. J Pediatr. 2009 May;154(5):700-7. doi: 10.1016/j.jpeds.2008.11.040. Epub 2009 Mar 4. PMID 19261295

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Part 1, subjects received Phenoptin for 8 days as part of their evaluation for Phenoptin responsiveness. Subjects who met response criteria were randomized 3:1 to Phenoptin or placebo for additional 10 weeks in Part 2, following a minimum 1-week wash-out period.
Period: Part 1: Responsiveness
Arm/Group | Sapropterin Dihydrochloride | Placebo
Started | 90 | 0
Completed | 89 | 0
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Part 2: Blinded, Placebo Control Period
Arm/Group | Sapropterin Dihydrochloride | Placebo
Started | 33 | 12
Completed | 32 | 9
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Patient Uncooperative | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sapropterin Dihydrochloride | Placebo | Total
Number analyzed (Participants) | 33 | 12 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (2.8) | 7.1 (2.0) | 7.5 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 20 | 6 | 26
Race [Number; unit: Participants]
  Caucasian | 33 | 11 | 44
  Hispanic | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Amount of Dietary Supplemented Phenylalanine (Phe)Tolerated in Children With Phenylketonuria
Time Frame: at Week 10
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Sapropterin Dihydrochloride | Placebo
Number analyzed (Participants) | 33 | 12
mg/kg/day | 20.9 (15.4) | 2.9 (4.0)
Statistical Analysis 1: Comparison: Sapropterin Dihydrochloride; Compared Week 10 to Baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided
Statistical Analysis 2: Comparison: Placebo; Compared Week 10 to Baseline; Test type: Superiority or Other; p = 0.027, t-test, 1 sided

2. Secondary Outcome: Change in Phenylalanine Levels From Baseline to Week 3
Time Frame: Baseline to Week 3
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Sapropterin Dihydrochloride | Placebo
Number analyzed (Participants) | 33 | 12
umol/L | -147.4 (29.0) | -90.3 (48.3)
Statistical Analysis 1: Comparison: Sapropterin Dihydrochloride vs Placebo; Test type: Superiority or Other; p = 0.009, Longitudinal Model; Longitudinal model with blood Phe measurements as the response variable and treatment group, visit, and baseline blood Phe level as covariates

ADVERSE EVENTS:
Arm/Group | Sapropterin Dihydrochloride | Placebo
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/12
Other Adverse Events (participants affected / at risk) | 26 | 8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Sapropterin Dihydrochloride | Placebo
Contusion (Injury, poisoning and procedural complications) | 3/33 (3) | 1/12 (1)
Excoriation (Injury, poisoning and procedural complications) | 2/33 (3) | 0/12 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0/33 (0) | 1/12 (1)
Streptococcal Infection (Infections and infestations) | 2/33 (2) | 2/12 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 2/33 (2) | 1/12 (1)
Appendicitis (Infections and infestations) | 0/33 (0) | 1/12 (1)
Conjuctivitis Infective (Infections and infestations) | 0/33 (0) | 1/12 (1)
Rhinitis (Infections and infestations) | 0/33 (0) | 1/12 (1)
Viral Infection (Infections and infestations) | 0/33 (0) | 1/12 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 7/33 (7) | 0/12 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5/33 (7) | 0/12 (0)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4/33 (5) | 1/12 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3/33 (4) | 0/12 (0)
Abdominal Pain (Gastrointestinal disorders) | 3/33 (6) | 1/12 (1)
Diarrhoea (Gastrointestinal disorders) | 4/33 (5) | 0/12 (0)
Vomiting (Gastrointestinal disorders) | 4/33 (4) | 0/12 (0)
Toothache (Gastrointestinal disorders) | 2/33 (2) | 0/12 (0)
Aphthous Stomatitis (Gastrointestinal disorders) | 0/33 (0) | 1/12 (1)
Headache (Nervous system disorders) | 7/33 (7) | 1/12 (1)
Rash (Skin and subcutaneous tissue disorders) | 1/33 (1) | 2/12 (4)
Erythema (Skin and subcutaneous tissue disorders) | 2/33 (2) | 0/12 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0/33 (0) | 1/12 (1)
Pyrexia (General disorders) | 3/33 (3) | 2/12 (2)
Fatigue (General disorders) | 1/33 (1) | 2/12 (2)
Neutrophil Count Decreased (Investigations) | 1/33 (1) | 1/12 (1)
White Blood Cell Count Decreased (Investigations) | 1/33 (1) | 1/12 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2/33 (2) | 0/12 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 2/33 (3) | 0/12 (0)
Depression (Psychiatric disorders) | 0/33 (0) | 1/12 (1)
Mood Swings (Psychiatric disorders) | 0/33 (0) | 1/12 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of the results shall be made by Sponsor in a joint publication. If such a multi-center publication is not submitted within 12 months after conclusion of the study, the PI may publish the results from their site individually, subject however to comply with the other terms of the agreement.